CLINICAL TRIAL: NCT04832919
Title: A Nurse-Community Health Worker-Family Partnership Model to Increase COVID19 Testing in Urban Underserved and Vulnerable Communities
Brief Title: A Nurse-Community Health Worker-Family Partnership Model: Addressing Uptake of COVID-19 Testing and Control Measures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3P30DA011041-23S1 (NIH)
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; COVID-19 testing; Behavioral COVID-19 Mitigation Measures
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Community Health Worker-Family Partnership (Experimental): The experimental arm will receive the Nurse-Community Health Worker-Family Partnership intervention
  Interventions: Behavioral: Nurse-Community-Family Partnership Intervention
- Standard of Care (No Intervention): The control arm will receive standard access to NYC Department of Health COVID-19 testing sites and standard COVID-19 public health messaging

INTERVENTIONS:
Behavioral: Nurse-Community-Family Partnership Intervention — Nurses conduct home visits on a monthly basis for the first five months post-baseline. During visits, nurses emphasize the importance of infection control measures and, jointly with household members, develop and follow-up on the implementation of an infection control plan tailored to the unique circumstances of the household. Nurses deliver training on infection control skills necessary for optimal implementation of the plan. Nurses offer at-home SARS-CoV-2 testing to all members of the household. Nurses conduct triage, medical case management, monitoring, and follow-up of individuals identified to have COVID-19 or any other acute health emergencies. CHWs conduct visits on a bi-weekly basis for the first five months post-baseline. CHWs deliver healthcare information and medical mistrust counseling in a culturally relevant and linguistically appropriate fashion; and provide social support, navigate household members to social welfare/vocational/economic/psychosocial services.
  Arms: Nurse-Community Health Worker-Family Partnership

SUMMARY:
Historically, health disparities in the US are concentrated among underserved communities and socially vulnerable populations. The disproportionate COVID-19 related morbidity and mortality in communities of color and socioeconomic disadvantage acutely highlight this persistent public health problem, drawing attention to the urgent need for more equitable reach of testing, prevention, and control measures. The proposed research addresses this need using a 2-arm randomized controlled trial (RCT) that will evaluate the effectiveness of the Nurse-Community Health Worker (CHW)-Family Partnership intervention in promoting COVID-19 testing uptake, adoption of COVID control measures, and mutual aid capacity at the household level in an underserved and vulnerable population disproportionately affected by COVID-19. Enrolled households will be randomly assigned to either the intervention group where families will receive the Nurse-CHW-Family Partnership intervention including the offer of in-home testing and referral to seasonal influenza vaccination services, or the treatment-as-usual control group, which will be used to measure actual testing rates among public housing residents in relation to participant and household characteristics. The study hypothesis is that the Nurse-CHW-Family Partnership intervention will improve household-level COVID-19 testing uptake, adoption of COVID control measures, and mutual aid capacity relative to the treatment-as-usual control.

DETAILED DESCRIPTION:
The investigators will recruit and follow a randomly-chosen sample of NYCHA public housing residents in the proposed target community who meet multiple criteria for being considered vulnerable or underserved. The current study will address knowledge gaps regarding COVID-19 testing, treatment, and household prevention strategies, and generate new knowledge related to the epidemiology of COVID-19 in these communities. Working with community partners, the investigators will create an acceptable and feasible intervention and testing infrastructure in advance of the influenza season, with a view toward designing best practices for sustainable COVID-19 testing, prevention, and preparedness for vaccination trials. The investigators will implement a 2-arm RCT that will evaluate the effectiveness of the Nurse-CHW-Family Partnership Intervention in promoting COVID testing uptake, adoption of COVID control measures, and household mutual aid capacity. The investigators will recruit members of randomly selected households in their homes using area sampling methods used with excellent results in the investigators' previous research in the target community. Participants will complete a baseline assessment and the entire household will be randomized to either the experimental or a treatment-as-usual control condition, which will be used to measure actual testing rates among public housing residents in relation to participant and household characteristics. The baseline sample will include 150 households, and 400 individual household members, randomized in a 2:1 ratio, intervention:control. Families will complete follow-up assessments at 6 and 9 months following the baseline. In-home testing and referral to seasonal influenza vaccination services will be offered to the intervention group; whereas the control group will receive treatment as usual at multiple NYC Department of Health COVID-19 testing sites that are within walking distance of each of the three housing complexes. Test acceptance will be recorded, and incentives will be paid for study visits, not for testing.

ELIGIBILITY:
Inclusion Criteria:

* Residence in one of the public housing complexes in Mott Haven, South Bronx
* English or Spanish-speaking
* Age 10 years or older
* Willing and able to provide informed consent or assent

Exclusion Criteria:

* Non-resident of one of the public housing complexes in Mott Haven, South Bronx
* Neither English nor Spanish speaker
* Younger than 10 years old, unless household index case tests antigen positive. In this instance, all members of family will be included.
* Unwilling or unable to provide informed consent or assent

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Household COVID-19 Testing Uptake | Delayed Follow-Up (9 Months)
  All medical services delivered by nurses during home-visits (such as COVID-19 test administration) will be carefully documented by the investigative team. At the time of the assessment, the investigators will obtain self-reported information regarding COVID-19 testing uptake by study participants in the treatment and control groups. Respondents will be asked whether they have received COVID-19 testing in the past three months [Yes/No].
COVID-19 Symptoms, Diagnoses, and Testing Scale | Delayed Follow-Up (9 Months)
  An adapted version of the (PhenX Toolkit) COVID-19 Symptoms, Diagnoses, and Testing Scale will be used to measure COVID-19 symptoms, diagnoses, and testing. Participants will be asked questions regarding whether they are currently sick with an illness that might be related to COVID-19, any symptoms the participant experienced in the past three months [Check All That Apply], and the result of the participant's last COVID-19 test [Positive/Negative].

SECONDARY OUTCOMES:
COVID-19 Avoidant Behaviors Scale | Delayed Follow-Up (9 Months)
  An adapted version of the COVID-19 Avoidant Behaviors Scale (PhenX Toolkit) will be used to measure the secondary study outcome of COVID-19 control measure uptake. Respondents will be asked questions regarding their engagement in behaviors associated with COVID-19 exposure on a 5-point scale [Almost Never, Sometimes, a Moderate Amount of the Time, Most of the Time, Always]; with greater values indicating higher frequency of uptake of COVID-19 prevention behaviors in the past three months (e.g., "Had close contact (within 6 feet) with people who do not live with you. "Gone out to a bar, club, or other place where people gather) and questions regarding their uptake of COVID-19 control (e.g., "Worn a mask or other face covering." "Washed your hands with soap or used hand sanitizer several times per day").
Vaccine Uptake | Delayed follow up (9 months)
  Referral to COVID-19 and seasonal influenza vaccination services by study nurses to intervention group participants will be carefully documented by the investigative team. At the time of the delayed assessment, the investigators will obtain self-reported information and documentation of COVID-19 and influenza vaccine uptake by study participants in the treatment as usual control group. For self-reported information, respondents will be asked if they received the flu shot in the past three months [Yes/No] and whether they received the COVID-19 vaccine [Yes/No], the type of vaccine, and the number of doses.
COVID-19 Improved Household & Family Mutual Aid | Delayed follow up (9 months)
  A set of measures will assess families' abilities to adjust to the COVID-19 pandemic, as evidenced by the reported overall impact of COVID-19 on family dynamics and relationships, psychological distress, food and housing insecurity, substance use, and sexual behavior in the past three months.
COVID-19 Household Environment Scale | Delayed follow up (9 months)
  An adapted version of the COVID-19 Household Environment Scale will be used to measure the secondary study outcome household/family mutual aid. The scale measures household conflict/togetherness. Participants are asked to rate, on a 5-point Likert scale, how much more or less conflict there was (as compared to before COVID-19) about 15 topics in the past three months (e.g., "Home maintenance;" "Decisions about visitors to the home"), with higher values indicating greater frequency of family conflict concerning the topic.
Household COVID-19 Testing Uptake | Immediate follow up (6 months)
  All medical services delivered by nurses during home-visits (such as COVID-19 test administration) will be carefully documented by the investigative team. At the time of the assessment, the investigators will obtain self-reported information regarding COVID-19 testing uptake by study participants in the treatment and control groups. Respondents will be asked whether they have received COVID-19 testing in the past six months [Yes/No].
COVID-19 Symptoms, Diagnoses, and Testing Scale | Immediate follow up (6 months)
  An adapted version of the (PhenX Toolkit) COVID-19 Symptoms, Diagnoses, and Testing Scale will be used to measure COVID-19 symptoms, diagnoses, and testing. Participants will be asked questions regarding whether they are currently sick with an illness that might be related to COVID-19, any symptoms the participant experienced in the past six months [Check All That Apply], and the result of the participant's last COVID-19 test [Positive/Negative].
COVID-19 Avoidant Behaviors Scale | Immediate follow up (6 months)
  An adapted version of the COVID-19 Avoidant Behaviors Scale (PhenX Toolkit) will be used to measure the secondary study outcome of COVID-19 control measure uptake. Respondents will be asked questions regarding their engagement in behaviors associated with COVID-19 exposure on a 5-point scale [Almost Never, Sometimes, a Moderate Amount of the Time, Most of the Time, Always]; with greater values indicating higher frequency of uptake of COVID-19 prevention behaviors in the past six months (e.g., "Had close contact (within 6 feet) with people who do not live with you. "Gone out to a bar, club, or other place where people gather) and questions regarding their uptake of COVID-19 control (e.g., "Worn a mask or other face covering." "Washed your hands with soap or used hand sanitizer several times per day").
Vaccine Uptake | Immediate follow up (6 months)
  Referral to COVID-19 and seasonal influenza vaccination services by study nurses to intervention group participants will be carefully documented by the investigative team. At the time of the assessment, the investigators will obtain self-reported information and documentation of COVID-19 and influenza vaccine uptake by study participants in the treatment as usual control group. For self-reported information, respondents will be asked if they received the flu shot in the past six months [Yes/No] and whether they received the COVID-19 vaccine [Yes/No], the type of vaccine, and the number of doses.
COVID-19 Improved Household & Family Mutual Aid | Immediate follow up (6 months)
  A set of measures will assess families' abilities to adjust to the COVID-19 pandemic, as evidenced by the reported overall impact of COVID-19 on family dynamics and relationships, psychological distress, food and housing insecurity, substance use, and sexual behavior in the past six months.
COVID-19 Household Environment Scale | Immediate follow up (6 months)
  An adapted version of the COVID-19 Household Environment Scale will be used to measure the secondary study outcome household/family mutual aid. The scale measures household conflict/togetherness. Participants are asked to rate, on a 5-point Likert scale, how much more or less conflict there was (as compared to before COVID-19) about 15 topics in the past six months (e.g., "Home maintenance;" "Decisions about visitors to the home"), with higher values indicating greater frequency of family conflict concerning the topic.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent M Guilamo-Ramos, PhD, Principal Investigator — New York University; Holly Hagan, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The project team will share all individual participant data that underlie the results reported in any future published manuscript, after deidentification (text, tables, figures, and appendices). We will make available the study protocol and statistical analysis plan. The project team will make the data available beginning 3 months and ending 5 years following article publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Investigators will be approved to conduct analyses to achieve the aims in the proposal that they submit for approval by an independent review committee. Proposals should be directed to Dr. Holly Hagan (hh50@nyu.edu). To gain access, data requesters will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: The project team will make the data available beginning 3 months and ending 5 years following article publication.
Access Criteria: The project team will make the data available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Guilamo-Ramos V, Benzekri A, Williams D, Thimm-Kaiser M, Wizentier MM, Goodman M, Amezquita-Castro B, Hagan H. A nurse-led clinical practice model to increase healthcare reach among underserved families during public health emergencies: A randomized controlled trial. Nurs Outlook. 2025 Nov-Dec;73(6):102591. doi: 10.1016/j.outlook.2025.102591. Epub 2025 Nov 6. PMID 41202466

DOCUMENTS (3):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT04832919/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT04832919/SAP_001.pdf
  • Informed Consent Form (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT04832919/ICF_002.pdf